CLINICAL TRIAL: NCT02899091
Title: A Randomized, Double-blind, Placebo-controlled, Phase I / IIa Clinical Trial for Evaluation of Safety and Potential Therapeutic Effect After Transplantation of CB-AC-02 in Patients With Alzheimer's Disease
Brief Title: Evaluation of the Safety and Potential Therapeutic Effects of CB-AC-02 in Patients With Alzheimer's Disease
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CHABiotech CO., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHA-PAD-101
Record Dates: First submitted 2016-09-02; First posted 2016-09-14 (Estimated); Last update posted 2024-04-09 (Actual); Status verified 2024-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Mesenchymal Stem cells
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CB-AC-02 (Experimental): Subjects with Alzheimer's disease Intervention: CB-AC-02
  Interventions: Biological: CB-AC-02
- Placebo (Placebo Comparator): Subjects with Alzheimer's disease Intervention: Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CB-AC-02 — Stage1:
  ① Group1: CB-AC-02 administration on day 0
  ② Group2: CB-AC-02 administration on day 0 and on week 4 (repeated injection)
  Stage2
  ① Arm1: K-MMSE 20~26 CB-AC-02 administration on day 0 and on week 4 (repeated injection)
  ② Arm2: K-MMSE 10~19 CB-AC-02 administration on day 0 and on week 4 (repeated injection)
  Arms: CB-AC-02
Biological: Placebo — Stage2:
  Placebo administration on day 0 and on week 4 (repeated injection)
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate safety and potential therapeutic effect of intraveneously administered CB-AC-02 in patients with Alzheimer's Disease.

DETAILED DESCRIPTION:
Subjects will receive either the single or multiple doses of CB-AC-02 to be followed up and evaluated for safety and potential therapeutic effect

ELIGIBILITY:
Inclusion Criteria:

1. Korean male or female at 50+ years of age at the time of screening visit
2. Diagnosis of Probable Alzheimer disease (probable AD) according to NINCDS-ADRDA criteria at Screening visit
3. Positive for Amyloid on amyloid-ligand PET
4. A subject with the imaging findings of Alzheimer's disease as confirmed by MRI or PET

   * Presence of brain atrophy on brain MRI by visual assessment
   * Presence of reduced brain glucose metabolism in bilateral temporal-parietal lobe on FDG-PET
5. Korea Mini-Mental State Examination (KMMSE) score of 10-26 at time of screening visit
6. Presence of caregiver who can provide information on the subject's condition
7. Subject who has been taking stable dose of Alzheimer medication for last 2 months or more
8. Subject who is informed of the clinical trial and signs a consent form (if unable to sign, a consent from a legally acceptable representative is required)

Exclusion Criteria:

1. Concurrent Dementia as a result of other disorders [i.e. infectious disease of the central nervous system such as HIV, syphilis, head injury, Creutzfeld-Jacob disease, Picks disease, Huntington's disease, Parkinson's disease, other subdural hematoma, hydrocephalus and structural brain lesions, drug addiction, alcoholism, substance abuse, thyroid disease, parathyroid disease, vitamins and other nutritional deficiencies and vascular etc.]
2. Subject with vascular dementia as determined by the clinical criteria of DSM-IV and the imaging criteria of Erkinkuntii
3. Subject with severe white matter hyperintensities (i.e. ≥ 25mm of the deep white matter and ≥ 10mm of the periventricular capping/banding in lengths)
4. Abnormal laboratory findings at screening visit
5. Subjects who are positive for HIV, syphilis or active HBV, HCV infection
6. Subjects in poor medical condition or subjects with severe cardiovascular, gastrointestinal, pulmonary or endocrinologic disease A. Suspected active active lung disease on chest X-ray at screening visit B. Diagnosis of cancer (except for the subjects who remains in complete remission for 5 years or more )
7. Subject with concurrent unstable psychiatric disorder (i.e. severe depression, or schizophrenia, or bipolar disorder, etc)
8. Pregnant or lactating women
9. Women of childbearing age who reject to practice contraception with one of the following methods

   * Use a condom
   * Use of contraceptive (oral, dermal, or injectable)
   * Use an intra-uterine contraceptive device
10. Subjects with a history of alcohol abuse (>30g/day) or drug abuse
11. Subjects who cannot undergo any of the tests performed in this clinical trial (for example, MRI, CT, PET, CSF study)
12. Subjects with known allergies to protein products (Bovine serum), antibiotics (gentamycin) or DMSO
13. Subjects whom the principal investigator considers inappropriate for participation in theis study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 48 weeks
  Number of subjects with treatment-related adverse events.
  The safety and tolerability of treatment with CB-AC-02 will be assessed by analysis of adverse events, abnormal findings on physical examinations, standard laboratory tests.

SECONDARY OUTCOMES:
Changes from the baseline in K-MMSE Score | 48 weeks
  K-MMSE, Korean-Mini Mental Status Examination
Change from the baseline of CMRglc analyzed with SPM (statistical parametric mapping) with Brain FDG PET imaging | 48 weeks
  CMRglc, cerebral metabolic rate for glucose
Changes from the baseline of Amyloid amount analyzed with SPM with amyloid PET imaging | 48 weeks
  SPM, statistical parametric mapping
Changes of band power in qEEG | 48 weeks
  qEEG, Quantitative electroencephalography

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Sook Kim, Principal Investigator — CHA University Bundang Medical Center
Locations (1):
- Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea